CLINICAL TRIAL: NCT05603104
Title: A Randomised, Controlled Trial to Investigate the Effect of an Intensified Pharmacological Treatment for Schizophrenia, Major Depressive Disorder and Bipolar Depression in Subjects Who Had a First-time Treatment Failure on Their First-line Treatment.
Brief Title: Intensified Pharmacological Treatment for Schizophrenia, Major Depressive Disorder and Bipolar Depression After a First-time Treatment Failure
Acronym: INTENSIFY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Inge Winter (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Sponsor-Investigator, Dr. Inge Winter, Workpackage leader, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-502185-24-00 (EU CT #)
Record Dates: First submitted 2022-10-13; First posted 2022-11-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia and Related Disorders; Major Depressive Disorder; Bipolar Depression
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder | interventions — Clozapine; Escitalopram; Sertraline; Venlafaxine Hydrochloride; Lithium; Quetiapine Fumarate; Ketamine; Bupropion

STUDY DESIGN:
Intervention Model Description: Parallel randomization to the treatment as usual (TAU) or early-intensified pharmacological treatment (EIPT) group for each of the study groups (schizophrenia, major depressive disorder, bipolar depression) leading to 6 arms.
Who Masked: Outcomes Assessor
Masking Description: Open label, except for the assesseors of the primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Schizophrenia EIPT: Switch to clozapine (Experimental): Schizophrenia randomized to EIPT: Switch to clozapine. Brand, dosage, frequency and duration up to the investigator's discretion
  Interventions: Drug: Clozapine
- Schizophrenia TAU: second-line antispychotic (Active Comparator): Schizophrenia randomized to TAU: switch to second-line antispychotic. Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC)
  Interventions: Drug: Second-line Antipsychotics
- Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray (Experimental): Major depressive disorder randomized to EIPT: Switch to second-line antidepressant + esketamine nasal spray or (es)ketamine infusion. Antidepressant: Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC).
  Esketamine nasal spray: 2 times per week for 4 weeks. Initial dose 28 mg, after that increases can be made with 28 mg per increase (up to 84 mg per week). This decision is up to the investigator's discretion (in accordance with SmPC).
  (Es)ketamine infusion: performed twice weekly for 4 weeks. Compound, brand up to the investigator's discretion (in accordance with SmPC).
  Interventions: Drug: Esketamine Nasal Product; Drug: Second-line Antidepressants; Drug: Ketamine Hydrochloride; Drug: Esketamine hydrochloride
- Major Depressive Disorder TAU: second-line antidepressant (Active Comparator): Major depressive disorder randomized to TAU: Switch to second-line antidepressant + esketamine nasal spray or ketamine IV or esketamine IV . Antidepressant: Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC).
  Interventions: Drug: Second-line Antidepressants
- Bipolar Depression EIPT: Switch to one of the following combinations: (Experimental): Bipolar Depression randomized to EIPT: Switch to 1. one of the following: escitalopram, sertraline, bupropion or venlafaxine plus 2. two of the following: lithium, valproate acid or quetiapine
  Interventions: Drug: Escitalopram; Drug: Sertraline; Drug: Venlafaxine; Drug: Lithium; Drug: Valproate acid; Drug: Quetiapine; Drug: Bupropion
- Bipolar Depression TAU: Switch to quetiapine plus lithium or valproate acid or lamotrigine (Active Comparator): Bipolar Depression randomized to TAU: Switch to quetiapine plus lithium or valproate acid Compound, brand, dosage, frequency and duration up to the investigator's discretion (in accordance with SmPC).
  Interventions: Drug: Lithium; Drug: Valproate acid; Drug: Quetiapine

INTERVENTIONS:
Drug: Clozapine — See arm description
  Other Names: ATC code: N05AH02
  Arms: Schizophrenia EIPT: Switch to clozapine
Drug: Esketamine Nasal Product — See arm description
  Other Names: ATC code: N06AB10
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray
Drug: Escitalopram — See arm description
  Other Names: ATC code: N06AB10
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:
Drug: Sertraline — See arm description
  Other Names: ATC code: N06AB06
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:
Drug: Venlafaxine — See arm description
  Other Names: ATC code: N06AX16
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:
Drug: Lithium — See arm description
  Other Names: ATC code: N05AN01
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:; Bipolar Depression TAU: Switch to quetiapine plus lithium or valproate acid or lamotrigine
Drug: Valproate acid — See arm description
  Other Names: ATC code: N03AG01
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:; Bipolar Depression TAU: Switch to quetiapine plus lithium or valproate acid or lamotrigine
Drug: Quetiapine — See arm description
  Other Names: ATC code: N05AH04
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:; Bipolar Depression TAU: Switch to quetiapine plus lithium or valproate acid or lamotrigine
Drug: Second-line Antidepressants — See arm description
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray; Major Depressive Disorder TAU: second-line antidepressant
Drug: Second-line Antipsychotics — See arm description
  Arms: Schizophrenia TAU: second-line antispychotic
Drug: Ketamine Hydrochloride — See arm description
  Other Names: N01AX03
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray
Drug: Esketamine hydrochloride — See arm description
  Other Names: N015X14
  Arms: Major Depressive Disorder EIPT: second-line antidepressant + esketamine nasal spray
Drug: Bupropion — See arm description
  Other Names: ATC code: N06AX12
  Arms: Bipolar Depression EIPT: Switch to one of the following combinations:

SUMMARY:
Schizophrenia, bipolar and major depressive disorders collectively affect over 10 million people across the EU and are associated with annual healthcare and societal costs in excess of 100 billion Euros. When diagnosed with one of these disorders, patients are prescribed psychotropic medication such as antidepressants, mood stabilisers or antipsychotics. It is unknown whether this first-line treatment will be successful. After this first-line treatment fails, usually a second-line treatment is initiated, and when this is not successful either a third-line treatment is initiated. Third-line treatments are quite successful, especially when compared to second-line treatments. The research question is whether the third-line treatments (early-intensified treatments) when used earlier in the disease course for schizophrenia, bipolar and major depressive disorders. If this is indeed the case, this could lead to the prevention of unnecessary trials of ineffective treatments and adaptations of worldwide guidelines as well as a reduction of healthcare and societal costs.

DETAILED DESCRIPTION:
Rationale Schizophrenia (SZ), bipolar depression (BD) and major depressive disorders (MDD) collectively affect over 10 million people across the European Union (EU) and are associated with annual healthcare and societal costs in excess of 100 billion Euros. When diagnosed with one of these disorders, patients are prescribed psychotropic medication such as antidepressants, mood stabilisers and/or antipsychotics. The effectiveness of these treatments for individual patients cannot be predicted. After this first-line treatment fails, usually a second-line treatment is initiated; when this is not effective either, a third-line treatment is initiated. Third-line treatments are quite effective, for people not responding to the first two treatments lines. However, they are used late in the disease course and clear evidence from direct comparisons of treatment algorithms is lacking. The research question is whether the third-line treatments would be more efficacious than the current second-line treatments (treatment as usual) for schizophrenia, bipolar and major depressive disorders. Third-line treatment can then be regarded as 'early-intensified'. If this is indeed the case, this could lead to the prevention of unnecessary trials of ineffective treatments and recommendations for adaptations of worldwide guidelines as well as a reduction of healthcare and societal costs. Additionally, The INTENSIFY trial is part of the larger Horizon 2021 project, with the central goal of paving the way for a shift towards a treatment decision-making process tailored for the individual at risk for treatment resistance. To that end, we aim to establish evidence-based criteria to make decisions of early intense treatment in individuals at risk for treatment resistance across the major psychiatric disorders of schizophrenia, bipolar disorder and major depression.

Objective The primary objective is to compare the treatment response, expressed as change in symptom severity as measured through the Positive And Negative Syndrome Scale (PANSS; SZ sample), and the Montgomery-Åsberg Depression Rating Scale (MADRS; MDD/BD samples) under an early-intensified pharmacological treatment to that under treatment as usual, in subjects who had a first-time treatment failure on their first-line treatment.

Main trial endpoints Change in symptom severity total score from baseline (visit 2) to end of treatment (visit 4). For SZ, this is measured using PANSS. For MDD and BD, MADRS is applied.

Secondary trial endpoints

1. All study samples: to compare changes in the severity and improvement sub-scores of the Clinical Global Impression Scale (CGI) between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
2. All study samples: to compare changes in the levels of depression and anxiety as assessed with the Hospital Anxiety and Depression Scale (HADS) between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
3. All study samples: to compare changes in cognitive performance as measured through the Trail Making Test, Digit Symbol Substitution Test, Rey Auditory Verbal Learning Test as well as the Perceived Deficits Questionnaire between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
4. All study samples: to compare changes in quality of life and functioning measures (Q-LES-Q-SF, LAPS, QLS-100 and SDS between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
5. All study samples: to compare presence of side effects as measured through General Assessment of Side Effects Scale (GASE) and reported spontaneously between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
6. All study samples: to compare use of concomitant medication between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
7. All study samples: to compare premature discontinuation (timing and reason)between the two treatment arms over the six week treatment period (visit 2 versus visit 4).
8. All study samples: comparison of the proportion of participants (EIPT vs. TAU) that is remission at visit 4. For SZ, remission is defined as meeting the PANSS modified Andreasen criteria (Low scores (≤3) P1. Delusions; P3. Hallucinatory behavior; P2. Conceptual disorganization; N1. Blunted affect; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity and flow of conversation; G5. Mannerisms/posturing; G9. Unusual thought content. For MDD/BD, remission is defined as a MADRS score ≤ 12
9. To compare changes in suicidal ideation between treatment arms.
10. SZ sample: to compare changes in PANSS subscale scores between the two treatment arms over the six-week treatment period (visit 2 versus visit 4).
11. BD study sample: To compare occurrence of (hypo)manic episode during the study between the treatment arms

Trial design The clinical study is an international, multicenter controlled, randomised, open label trial, with a treatment duration of 6 weeks.

Trial population The aim is to recruit 418 subjects into each of the study samples, leading to a total sample size of 1254 subjects. The study samples are: schizophrenia (schizophrenia, schizoaffective disorder or schizophreniform disorder), major depressive disorder and bipolar depressive disorder (bipolar I or II disorder currently in a depressive episode). Male and female subjects, in- and out-patients, within the age of at least 18 years old are eligible for participation. The main exclusion criteria to protect the subjects are subjects being pregnant or breastfeeding, subjects with previous failure on the early-intensified pharmacological treatments, known intolerance to any of the treatments or meeting any contraindications for the early-intensified pharmacological treatments.

Interventions

Per study sample (SZ, MDD, BD), subjects are randomised to treatment as usual (second-line treatment) or to the early-intensified pharmacological treatment (third-line treatment). Treatment per group per study sample can be found below:

SZ sample:

Treatment as Usual (TAU): Switch to second line antipsychotic Early-Intensified Pharmacological Treatment (EIPT): Switch to clozapine

MDD sample:

Treatment as Usual (TAU): Switch to second-line antidepressant Early-Intensified Pharmacological Treatment (EIPT): Oral antidepressant plus esketamine nasal spray or esketamine IV or ketamine IV

BD sample:

Treatment as Usual (TAU): Switch to quetiapine plus lithium or valproate acid

Early-Intensified Pharmacological Treatment (EIPT): Switch to:

1. one of the following: escitalopram, sertraline, bupropion or venlafaxine plus
2. two of the following: lithium, valproate acid or quetiapine

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of subjects represented by the trial subjects as well as the nature and extent of burden and risks All medications studied in the current trial are widely used (alone or in combination) in clinical practice and the risks for side effects are well established. In the current study, clinical practice is mimicked as much as possible to maximize generalizability and for feasibility purposes. To this end, Summaries of Product Characteristics (SmPCs) are followed with regards to contraindications (implemented as exclusion criterion), safety measures and allowed combinations with other medications. Site visits and assessments are kept to a minimum to keep subject burden at an acceptable level, while meeting the objectives of the study. Blood samples are only collected when subjects provide consent; safety measures are performed as part of clinical routine.

Overall, the risks are similar to daily clinical practice; the only difference relative to clinical practice is the application of early-intensified pharmacological treatment earlier in the illness. However, these intense treatment options are also commonly prescribed by clinicians. There are no indications in existing literature that the earlier introduction of these medications poses a safety risk.

A benefit of the study is that if it indeed turns out that the early-intensified pharmacological treatment is associated with more symptom improvement compared to treatment as usual, treatment guidelines may be changed accordingly and early-intensified pharmacological treatment becomes available earlier in the illness course, as second-line treatment. This would mean that future subjects have to go through less trial and error, which results in a reduced burden for subjects as well as lower societal and healthcare costs.

IMPORTANT: the study was submitted to the European suthorities and they requested to split this study into 3 studies (1 for each diagnostic category). We have done this and created 3 new ClinicalTrials.gov studies as well. The numbers are NCT05958875 (SZ substudy), NCT05973786 (BD substudy) and NCT05973851 (MDD substudy).

The site in the UK (London) followed the advice and will submit 3 separate protocols. However, Israel already submitted this as one protocol. Therefore, we keep this clinicaltrials.gov number for Israel.

ELIGIBILITY:
Inclusion Criteria:

1. In- or out patients, at least 18 years of age up until 70 (SZ study sample), 65 years (MDD study sample) and no limit for the BD study..

Being willing and able to provide written informed consent. Having a legal guardian to cosign is allowed. Informed consent will be signed at visit 1, before any study procedure.

3. Female subjects of child bearing potential must be willing to ensure that they use effective contraception during the trial and as per the requirements in the protocol (section 8.2.1).Male subjects that will use valproate acid during the trial must use effective contraceptive measures during the trial.

4. Meeting diagnostic criteria for a primary diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, major depressive disorder (without psychotic features) or bipolar depression (bipolar disorder type I and II currently in a depressive episode), according to DSM-5. The primary diagnosis will be confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2).

5. Subject experiences a treatment failure due to lack of efficacy in the current episode, as confirmed by a CGI-I ≥3; preferably this treatment is a first-line pharmacotherapeutic agent for the primary DSM-5 diagnosis, and was prescribed for at least 4 weeks within an effective dose range as specified in the Summary of Product Characteristics (SmPCs). However, other lines of treatment are accepted as well.

6. Subject and clinician intend to change pharmacotherapeutic treatment. 7. A minimum symptom severity threshold needs to be present (moderate level; see below) and subject needs to experience functional impairment.

* The minimum symptom severity threshold for SZ subjects is at least 2 PANSS positive or negative items with a score of 4, or at least one PANSS positive or negative item with a score of 5.
* The minimum symptom severity threshold for MDD is a score of ≥ 20 on the Montgomery Åsberg Depression Rating Scale (MADRS)
* The minimum symptom severity threshold for BD is a score of ≥20 on the Montgomery Åsberg Depression Rating Scale (MADRS)
* For all study samples: Functional impairment is defined as a score of 5 or higher on any of the three scales of the Sheehan Disability Scale (SDS).

Exclusion criteria:

1. Being pregnant or breastfeeding.
2. Subject has failed previously on the EIPT study medication (i.e. SZ: clozapine; MDD: esketamine intranasal/(es)ketamine IV) Treatment duration as ≥ 4 weeks within an efficacious dose range according to the SmPC.
3. Subject has a known intolerance to clozapine (SZ only), esketamine intranasal/ (es)ketamine IV (MDD only) or quetiapine (BD only) or to all medication options for a study sample (related to the TAU treatment arms) or all EIPT medications (BD study sample).
4. Meeting any of the contraindications of clozapine (SZ only), esketamine intranasal/ (es)ketamine IV (MDD only) or quetiapine (BD only), or to all medication options for a study sample (related to the TAU treatment arms), or all EIPT medications (BD study sample), as specified within the applicable SmPC.
5. Subject has participated in another clinical trial in which the subject received an experimental or investigational drug or agent within 30 days before visit 1.
6. Subject experiences any other significant disease or disorder which, in the opinion of the investigator, may either put the subjects at risk because of participation in the trial, or may influence the result of the trial, or the subject's ability to participate in the trial.
7. 7. Subjects with active suicidal ideation with some intent to act, without specific plan ("Yes" to question 4 of the Columbia-Suicide Severity Rating Scale (C-SSRS)) or active suicidal ideation with specific plan and intent ("Yes" to question 5 of the C-SSRS), followed by an assessment by the treating clinician who determines it is not safe for the subject to participate in the study
8. Subject meets criteria for current substance use disorder, as confirmed by the Mini International Neuropsychiatric Interview (MINI v7.0.2). Nicotine dependency is allowed, as well as mild and moderate alcohol and/or cannabis use disorder (as defined by MINI v7.0.2). Severe alcohol and/or cannabis use disorder are not allowed.
9. Subjects have not been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
10. Subjects dependent on the sponsor, investigator or trial site must be excluded from participation in advance.
11. For the SZ sample only: schizophrenia subjects cannot meet the modified Andreasen criteria for remission.
12. For the SZ sample only: Subjects that have any clinically significant abnormal values on the local laboratory test (especially ANC/WBC and liver values), electrocardiogram (ECG) or physician examinations.
13. For the BD sample only: a score of 12 or higher on the Young Mania Rating Scale (YMRS) in order to exclude subjects with predominant manic symptoms or mixed symptoms.
14. For the BD study sample only: Subjects with a history of antidepressant-induced mania or hypomania or recent rapid cycling (based on the medical file of the potential participant or the clinical judgment of the clinician).
15. For the BD study sample only: Subjects with pre-existing severe liver damage (as tested within the local laboratory test at visit 1).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity | 6 weeks
  Change in symptom severity total score from baseline (visit 2) to end of treatment (visit 4). For Schizophrenia, this is measured using the Positive And Negative Syndrome Scale. For Major Depressive Disorder and Bipolar Depression, Montgomery Åsberg Depression Rating Scale is applied.

SECONDARY OUTCOMES:
All study samples: to compare changes in the severity and improvement | 6 weeks
  All study samples: to compare changes in the severity and improvement sub-scores of the Clinical Global Impression Scale between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare changes in the levels of depression and anxiety | 6 weeks
  All study samples: to compare changes in the levels of depression and anxiety as assessed with the Hospital Anxiety and Depression Scale bbetween the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare changes in cognitive performance #1 | 6 weeks
  All study samples: to compare changes in cognitive performance as measured through the Trail Making Test between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare changes in cognitive performance #2 | 6 weeks
  All study samples: to compare changes in cognitive performance as measured through the Digit Symbol Substitution Test between the two treatment arms over four weeks (Major Depressive Disorder Group)/six weeks (Schizophrenia/Bipolar Depression groups) treatment period (visit 2 versus visit 4).
All study samples: to compare changes in cognitive performance #3 | 6 weeks
  All study samples: to compare changes in cognitive performance as measured through the Rey Auditory Verbal Learning Test between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare changes in cognitive performance #4 | 6 weeks
  All study samples: to compare changes in cognitive performance as measured through the Perceived Deficits Questionnaire between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare changes in functioning measure #1 | 6 weeks
  All study samples: to compare changes in functioning measure (Leuven Afective and Pleasure Scale) between the two treatment arms over the four weeks (Major Depressive Disorder Group)/six weeks (Schizophrenia/Bipolar Depression groups) treatment period (visit 2 versus visit 4).
All study samples: to compare changes in functioning measure #2 | 6 weeks
  All study samples: to compare changes in functioning measure (Sheehan Disability Scale) between the two treatment arms over the four weeks (Major Depressive Disorder Group)/six weeks (Schizophrenia/Bipolar Depression groups) treatment period (visit 2 versus visit 4).
All study samples: to compare changes in quality of life #1 | 6 weeks
  All study samples: to compare changes in quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire Short Form) between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare changes in quality of life #2 | 6 weeks
  All study samples: to compare changes in quality of life and functioning measures (Quality of Life Scale -100, subscale inner tension) between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare presence of side effects | 6 weeks
  All study samples: to compare presence of side effects as measured through General Assessment of Side Effect Scale between the two treatment arms over the two treatment arms over the four weeks (Major Depressive Disorder Group)/six weeks (Schizophrenia/Bipolar Depression groups) treatment period (visit 2 versus visit 4).
All study samples: to compare use of concomitant medication | 6 weeks
  All study samples: to compare use of concomitant medication between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: to compare premature treatment discontinuation | 6 weeks
  All study samples: to compare premature treatment discontinuation (timing and reason) between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
Schizophrenia sample: to compare changes in Positive and Negative syndrome subscale scores | 6 weeks
  Schizophrenia sample: to compare changes in Positive and Negative syndrome subscale scores between the two treatment arms over the six weeks treatment period (visit 2 versus visit 4).
All study samples: comparison of the proportion of participants (EIPT vs. TAU) that is remission at visit 4. | 6 weeks
  For SZ, remission is defined as meeting the PANSS modified Andreasen criteria (Low scores (≤3) P1. Delusions; P3. Hallucinatory behavior; P2. Conceptual disorganization; N1. Blunted affect; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity and flow of conversation; G5. Mannerisms/posturing; G9. Unusual thought content. For MDD/BD, remission is defined as a MADRS score ≤ 12
All study samples: To compare changes in suicidal ideation between treatment arms. | 6 weeks
  Changes on the Columbia-Suicide Severity Rating Scale (C-SSRS) throughout the study; EIPT vs TAU. Higher scores means higher suicidal ideation. The maximum score is 5.
BD study sample: To compare occurrence of (hypo)manic episode during the study between the treatment arms using the Young Mania Rating Scale | 6 weeks.
  Occurrence of (hypo)manic episodes throughout the study (including V5); EIPT vs TAU. Scores of 12 or higher means that a participant is in a (hypo)manic episode of bipolar disorder.
  The minimum score on the YMRS is 0 and the maximum score 60.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR